CLINICAL TRIAL: NCT03701607
Title: Effect of Platinum-based Chemotherapy on PD-L1 Expression in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Effect of Chemotherapy on PD-L1 in NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baodong Qin (Other)
Responsible Party: Sponsor-Investigator, Baodong Qin, Principal Investigator, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Other Study IDs: COPDL1
Record Dates: First submitted 2018-09-16; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Chemotherapy; Immunotherapy; PD-L1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PD-L1
  Interventions: Other: PD-L1 group

INTERVENTIONS:
Other: PD-L1 group — PD-L1 expression is evaluated using immunohistochemical assay

SUMMARY:
PD-L1 is identified as an important biomarkers for predicting PD-1/PD-L1 inhibitors in advanced Non-Small Cell Lung Cancer. Several previous clinical trials have demonstrated that chemotherapy could enhance the efficacy of PD-1/L1 immunotherapy in NSCLC such as Checkmate-227, Impower-150, Keynote-189, etc. Pre-clincial experiment shows that chemotherapy could increase CD8 TIL infiltration in tumor microenvironment, activate T cell immune reaction. However, it remains unclear whether chemotherapy could affect PD-L1 in advanced NSCLC patients. The present study aims to evaluate whether PD-L1 will change after receiving chemotherapy in advanced NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC diagnosed histologically; Expected survival ≥ 6 month;
* Without Druggable molecular events (EGFR, ALK, c-Met, BRAF, Ret, etc)
* ECOG / PS score: 0-2, and the main organ function to meet the following criteria: HB ≥ 90g / L, ANC ≥ 1.5 × 109 / L, PLT ≥ 80 × 109 / L,BIL <1.5 times the upper limit of normal (ULN); Liver ALT and AST <2.5 × ULN and if liver metastases, ALT and AST <5 × ULN; Serum Cr ≤ 1 × ULN, endogenous creatinine clearance ≥50ml/min

Exclusion Criteria:

* Patient can not comply with research program requirements or follow-up;
* Patient will receive immunotherapy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced NSCLC without druggable molecular events (EGFR, ALK, c-Met, BRAF, Ret, etc)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with PD-L1 positive as assessed by immunohistochemical assay | through study completion, an average of 1 year
  PD-L1 will be calculated using immunohistochemical assay

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No